CLINICAL TRIAL: NCT00460057
Title: The Change of Bone Markers After Low Dose Alendronate in Postmenopausal Women
Brief Title: The Change of Bone Markers After Low Dose Alendronate in Postmenopausal Women With Bone Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eulji University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Jeong Choi, Associate Professor, Eulji University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EJRG-06-001-11E32
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Osteoporosis
Keywords: osteoporosis; alendronate; bone marker
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Diphosphonates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alendronate, Placebo (Placebo Comparator): All subjects were given 600 mg of calcium and 400 IU of vitamin D supplements. The subjects were randomized to receive weekly alendronate 20 mg (n = 31) or placebo (n = 32).
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Take two tablets (alendronate 10 mg) once weekly with a full glass of plain water in the morning after an overnight fast and to refrain from lying down or taking any other beverage or food for at least 1 h thereafter
  Other Names: Bisphosphonate

SUMMARY:
High bone turnover with the bone resorption exceeding bone formation is a major mechanism of postmenopausal osteoporosis. Therefore, inhibition of bone resorption is a rational approach for the prevention. The Objective of the current study was to determine the short-term efficacy of once-weekly low dose alendronate in the prevention of bone loss in early postmenopausal Korean women with moderate bone loss via bone turnover markers.

This study was a 12-week, randomized, double-blind clinical trial compared the effects of placebo with alendronate 20 mg once weekly. All subjects received supplemental calcium 600 mg and vitamin D 400 IU daily. Fifty two postmenopausal women (the ages between 50-65 year) with lumbar spine BMD at least 2.0 SD below the peak young adult mean were recruited at Eulji University Hospital, Daejeon, Korea. BMD was measured by DXA at baseline and serum alkaline phosphatase, osteocalcin and C-terminal telopeptide of type I collagen was measured at baseline and 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women (the ages between 50-65 year) with lumbar spine BMD at least 2.0 SD below the peak young adult mean

Exclusion Criteria:

* severe osteoporosis
* current medication of osteoposis
* metabolic bone disease
* cancer, stroke etc.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Changes of bone turnover markers | 12 weeks
  to determine the short-term efficacy of once-weekly low-dose alendronate, via bone turnover markers and OPG, in the prevention of bone loss in early postmenopausal Korean women with moderate bone loss.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Jeong Choi, MD, PhD, Principal Investigator — Department of Family medicine, Eulji University Hospital